CLINICAL TRIAL: NCT00397982
Title: A Phase II Study of CCI-779 in Combination With Bevacizumab in Stage III or IV Melanoma
Brief Title: Temsirolimus and Bevacizumab in Treating Patients With Stage III or Stage IV Malignant Melanoma
Acronym: Mel47
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00133; NCI-2009-00133 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-7190; CDR0000512836; UVACC-MEL-47; MEL47 (Other: University of Virginia Cancer Center); 7190 (Other: CTEP); P30CA044579 (NIH); R21CA128367 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Recurrent Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor, monoclonal antibody) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1 and 8 and bevacizumab IV over 30-90 minutes on day 8. Treatment repeats every 14 days for a maximum of 26 courses in the absence of disease progression or unacceptable toxicity. Patients undergo tumor resection on day 9 of course 2.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Temsirolimus; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
Procedure: Therapeutic Conventional Surgery — Undergo tumor resection

SUMMARY:
This phase II trial is studying how well giving temsirolimus together with bevacizumab works in treating patients with stage III or stage IV malignant melanoma. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of malignant melanoma by blocking blood flow to the tumor. Giving temsirolimus together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective tumor response rate (complete response and partial response) in patients with stage III or IV melanoma treated with temsirolimus and bevacizumab.

SECONDARY OBJECTIVES:

I. Describe the adverse event profile of this regimen in these patients. II. Determine the efficacy of this regimen, in terms of progression-free survival, in these patients.

III. Compare pre- vs post-treatment measurements of biomarkers and vascular system/immune system parameters in patients treated with this regimen.

IV. Correlate tumor and blood biomarkers with clinical response in these patients.

OUTLINE: This is a multicenter study.

Patients receive temsirolimus intravenously (IV) over 30 minutes on days 1 and 8 and bevacizumab IV over 30-90 minutes on day 8. Treatment repeats every 14 days for a maximum of 26 courses in the absence of disease progression or unacceptable toxicity. Patients undergo tumor resection on day 9 of course 2.Blood samples are collected during courses 1 and 2. Samples are examined by flow cytometry to evaluate peripheral blood mononuclear cells for molecular effects of study agents. Patients also undergo normal and tumor tissue biopsy (by core needle biopsy, incisional biopsy, or surgical resection) during courses 1 and 2. Samples are examined by immunohistochemistry, western blotting, protein array technology, gene expression analyses, DNA mutation analyses, and genomic analyses for pre-and post-treatment measurements of target molecules (epidermal growth factor receptor, B-Raf, MEK, MAPK), downstream pathway components (PI-3 kinase, AKT, mTOR), markers of angiogenesis, proliferation and apoptosis, markers that may modulate cell signaling or the response to investigational agents, and vascular and immune system parameters.

After completion of study treatment, patients are followed at 1 month, every 3 months for up to 2 years, and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma

  * Stage III or IV disease

    * Recurrent disease allowed
* Measurable disease defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm with conventional techniques OR ≥ 10 mm with spiral CT scan

  * Tumor lesions in previously irradiated areas are not considered measurable disease
* Prior brain metastases allowed provided all of the following criteria are met:

  * No more than a total of 5 brain metastases
  * All metastases are no more than 2.5 cm
  * Surgically resected or have been treated with gamma-knife or stereotactic radiosurgery
  * More than 30 days since prior disease progression
  * More than 30 days since prior steroids for managing brain metastases

    * Concurrent steroids for other reasons allowed provided the dose is < that required for managing brain metastases
* Disease accessible for core needle biopsy, incisional biopsy, and/or surgical resection and meets one of the following criteria:

  * One large tumor deposit ≥ 5 cm³ from which biopsies can be harvested multiple times
  * Multiple deposits that can be biopsied or excised individually on different dates, measured as follows:

    * One lesion ≥ 5 cm^3
    * Two lesions ≥ 3 cm^3
    * Three lesions ≥ 2 cm^3
* ECOG performance status 0-1
* Weight ≥ 110 pounds (without clothes)
* WBC ≥ 3,000 mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Urine protein: creatinine ratio < 1.0 OR 24-hour urine protein < 1,000 mg
* Fasting cholesterol < 350 mg/dL (cholesterol medications are allowed)
* Fasting triglycerides < 400 mg/dL
* PT INR ≤ 1.5 (unless on full-dose anticoagulants)
* Hematocrit < 41% (for males) or < 38% (for females)
* None of the following within the past 4 weeks:

  * Uncontrolled intercurrent illness
  * Ongoing or active acute (CTCAE v.3 grade 3 or 4) infection
  * Abdominal fistula
  * Gastrointestinal perforation
  * Intra-abdominal abscess
  * Serious or nonhealing wound, ulcer, or bone fracture
* No psychiatric illness or social situations that would preclude study compliance
* No clinically significant cardiovascular disease, including the following:

  * Cerebrovascular accident within the past 6 months
  * Transient ischemic attack within the past 6 months
  * Myocardial ischemia within the past 6 months
  * Myocardial infarction within the past 6 months
  * Other thromboembolic event within the past 6 months
  * Unstable angina within the past 6 months
  * Uncontrolled hypertension (i.e., hypertension despite maximal therapy)
  * New York Heart Association class II-IV heart disease
  * Congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Clinically significant peripheral vascular disease
  * History of stroke
  * Artificial valve, pacemaker, or similar device
* No uncontrolled diabetes

  * Hemoglobin A1c < 7%
* No significant traumatic injury within the past 28 days
* No history of allergic reactions to compounds of similar chemical or biological composition to temsirolimus or bevacizumab
* No hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies (e.g., infliximab)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* HIV negative
* Hepatitis C negative
* See Disease Characteristics
* More than 4 weeks since any of the following prior treatments and recovered:

  * Chemotherapy (6 weeks for nitrosoureas or mitomycin C)
  * Radiotherapy to nontarget lesions or lesions that are not to be biopsied
  * Immunotherapy
  * Cytokine therapy
  * Enzyme-inducing antiepileptic drugs (EIAEDs) or other CYP3A4 inducers
  * Investigational agents
* More than 4 weeks since prior major surgery or open biopsy and recovered
* No prior temsirolimus, rapamycin, bevacizumab, or systemic therapies targeted primarily to vascular endothelial growth factor (VEGF), VEGF receptors, or to mTOR inhibition
* Concurrent full-dose anticoagulants (e.g., warfarin/low molecular weight heparin) with PT INR > 1.5 are allowed provided the following criteria are met:

  * In-range INR (usually between 2 and 3.5) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * No active, clinically significant bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)

    * Minimal tumor bleeding of the skin allowed at the clinician's discretion
* No concurrent medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of the following:

  * Temsirolimus
  * Bevacizumab
  * CYP450 isoenzymes
* No concurrent nonstudy-related surgical procedures
* No other concurrent anticancer agents or therapies

Exclusion Criteria

* Participants who have received these medications or treatments at any time ≤ 4 weeks of registration:

  * Chemotherapy
  * Radiotherapy to non-target lesions and lesions that are not to be biopsied. Prior radiotherapy to target lesions or lesions to be biopsied/resected is not permitted
  * Immunotherapy
  * Cytokine therapy
  * Investigational reagents
  * Invasive procedures defined as follows:

    * Major surgical procedure, open biopsy or significant traumatic injury
    * Anticipation of need for non-study related surgical procedures from registration until Cycle 26 (One year).
  * Enzyme-inducing antiepileptic drugs (EIAEDs) or any other CYP3A4 inducer (Appendix C).

OR Participants who have not recovered from adverse events resulting from the administration of these agents/procedures > 4 weeks prior to registration.

* Participants who have received nitrosureas or mitomycin C ≤ 6 weeks of registration.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CCI-779 or bevacizumab, or with known hypersensitivity to Chinese hamster ovary cell products (t-PA) or other recombinant human antibodies (e.g., Remicade®).
* Participants who have previously received CCI-779, rapamycin, bevacizumab, or systemic therapies targeted primarily to VEGF, VEGF receptors, or to mTOR inhibition.
* Participants who have experienced any of the following ≤ 4 weeks prior to registration:

  * Uncontrolled intercurrent illness
  * Infection, CTCAE3 grade 3 or 4 (either ongoing, chronic, or active infection)
  * Abdominal fistula
  * Gastrointestinal perforation
  * Intra-abdominal abscess
  * Serious or non-healing wound
  * Serious or non-healing ulcer
  * Serious or non-healing bone fracture.
* Potential subjects with clinically significant cardiovascular disease

  * Recent history (defined as ≤ 6 months of registration) of thromboembolic events including cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial ischemia, myocardial infarction (MI)
  * Uncontrolled hypertension (hypertension despite maximal therapy)
  * Unstable angina ≤ 6 months of registration
  * New York Heart Association Classification of ≥ class II heart disease
  * Congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Clinically significant peripheral vascular disease
  * Have a history of stroke
  * Have an artificial valve, pace-maker, or similar device
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant (positive pregnancy test) or nursing women. Both fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of their participation in the study therapy.
* PT INR > 1.5, (unless the potential subject is on full dose anticoagulants and meet criteria described in Section 3.1.8).
* Participants with uncontrolled diabetes, defined as having a HGBA1C ≥ 7%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Slingluff, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Slingluff CL Jr, Petroni GR, Molhoek KR, Brautigan DL, Chianese-Bullock KA, Shada AL, Smolkin ME, Olson WC, Gaucher A, Chase CM, Grosh WW, Weiss GR, Wagenseller AG, Olszanski AJ, Martin L, Shea SM, Erdag G, Ram P, Gershenwald JE, Weber MJ. Clinical activity and safety of combination therapy with temsirolimus and bevacizumab for advanced melanoma: a phase II trial (CTEP 7190/Mel47). Clin Cancer Res. 2013 Jul 1;19(13):3611-20. doi: 10.1158/1078-0432.CCR-12-3919. Epub 2013 Apr 25. PMID 23620404
- [Result] Wagenseller AG, Shada A, D'Auria KM, Murphy C, Sun D, Molhoek KR, Papin JA, Dutta A, Slingluff CL Jr. MicroRNAs induced in melanoma treated with combination targeted therapy of Temsirolimus and Bevacizumab. J Transl Med. 2013 Sep 18;11:218. doi: 10.1186/1479-5876-11-218. PMID 24047116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from Jan 2008 - Feb 2011 at the University of Virginia Cancer Center and Fox Chase Cancer Center.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody)
Started | 17
Completed | 13
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — noncompliance | 1
Not completed — Unrelated health issues | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study: Patients receive temsirolimus IV over 30 minutes on days 1 and 8 and bevacizumab IV over 30-90 minutes on day 8. Treatment repeats every 14 days for a maximum of 26 courses in the absence of disease progression or unacceptable toxicity. Patients undergo tumor resection on day 9 of course 2.
  Bevacizumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV
  Therapeutic Conventional Surgery: Undergo tumor resection
Arm/Group | Entire Study
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response (Complete Response and Partial Response) and Progression in Participants With Stage III or IV Melanoma Following Treatment With Temsirolimus and Bevacizumab
Description: Evaluated using Response Evaluation Criteria In Solid Tumor (RECIST) criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: Up to 18 weeks after registration.
Measure: Number; unit: participants
Groups:
- Entire Study: Treatment
Arm/Group | Entire Study
Number analyzed (Participants) | 17
participants
  Partial response | 3
  Stable disease at 8 weeks | 9
  Progressive disease | 4
  not evaluable | 1

2. Secondary Outcome: Adverse Events in Participants With Stage III or IV Melanoma Treated With Temsirolimus and Bevacizumab
Description: Defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome, or disease which either occurs during the study (having been absent at baseline) or if present at baseline, appears to worsen. Graded using scales found in the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Tabulated by type and severity: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: On days 1 and 8 of each cycle, and up to 2 years after registration.
Population: Treatment related adverse events.
Measure: Number; unit: participants
Groups:
- Entire Study: 17 participants
Arm/Group | Entire Study
Number analyzed (Participants) | 17
participants
  grade 3 hypokalemia | 2
  grade 3 hypophosphatemia | 2
  grade 3 weight loss | 2
  grade 4 lymphopenia | 2
  grade 2 leukoencephalopathy | 1

3. Secondary Outcome: Association Between Expression or Activation of One Biomarker With Another, With Biochemical and Clinical Responses, With Alterations in Cell Proliferation and Apoptotic Markers, and With Time to Progression
Description: Changes in the ratio of phospho-S6Kinase (pS6K) S240/244 to total S6, in the tumor, from day 1 to day 23. These were assessed by reverse-phase protein array. A linear model was fit with PROC MIXED in SAS 9.3 using the log base 10 of expression as the outcome measure. This measure type is not listed in the data table form; so the number of patients who had decreases in that ratio is listed.
Time Frame: Day 1 of course 1 and day 8 of course 2
Population: This analysis was performed for those participants with sufficient tumor available for analysis.
Measure: Number; unit: participants who had decreases in ratio
Arm/Group | Entire Study
Number analyzed (Participants) | 13
participants who had decreases in ratio | 13

4. Secondary Outcome: Comparison of Biomarkers to Antitumor Activity/Patient Outcomes
Description: Assessed in both tumor tissue pretreatment. Mutations in BRAF were assessed in all 16 of the patients and were assessed for any association with clinical response
Time Frame: Day 1 of course 1 and day 8 of course 2
Population: Patients evaluable for clinical outcome with BRAF mutation status.
Measure: Count of Participants; unit: Participants
Arm/Group | Entire Study
Number analyzed (Participants) | 16
Participants
  BRAF-wild type: number analyzed (Participants) | 10
  BRAF-wild type: Partial responses | 3
  BRAF-wild type: Stable disease at 8 wks | 5
  BRAF-wild type: Progressive disease | 2
  BRAF-mutant: number analyzed (Participants) | 6
  BRAF-mutant: Partial responses | 0
  BRAF-mutant: Stable disease at 8 wks | 4
  BRAF-mutant: Progressive disease | 2

5. Secondary Outcome: Comparison of Pre- vs Post-treatment Measurements of Biomarkers and Vascular System/Immune System Parameters
Description: Biomarker expression in tumor and normal skin will be assessed by immunohistochemistry (IHC) or Western blotting, using marker-specific antibodies.
Time Frame: Day 1 of course 1 and day 8 of course 2
Population: Detailed vascular changes were not assessed.
Arm/Group | Entire Study
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-free Survival
Description: Defined as the duration of time from start of treatment to time of progression, death or date of last follow-up.
Time Frame: Day 11 of courses 4, 8, 12, 16, 20, and 24, and then annually for up to 5 years
Population: Entire study
Measure: Median (Full Range); unit: months
Arm/Group | Entire Study
Number analyzed (Participants) | 17
months | 4.6 [1.1 to 32.7]

ADVERSE EVENTS:
Time Frame: Up to 2 years after registration
Description: CTCAE 3.0.
Arm/Group | Entire Study
Serious Adverse Events (participants affected / at risk) | 9/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study (N=17)
Leukoencephalopathy (Nervous system disorders) | 1 (1) — grade 2 leukoencephalopathy, reversible.
lymphopenia (Blood and lymphatic system disorders) | 2 (2) — grade 4 lymphopenia, both were evident pre-treatment at grade 1 and grade 3 for the two patients, respectively.
lymphopenia (Blood and lymphatic system disorders) | 1 (1) — grade 3 lymphopenia
hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) — grade 3
Anemia (Blood and lymphatic system disorders) | 1 (1) — grade 3 anemia (hemoglobin)
Opportunistic infection (Infections and infestations) | 1 (1) — grade 3
Hypertension (Cardiac disorders) | 1 (1) — grade 3 hypertension
Mucositis (funct/sympt) - Oral cavity (Gastrointestinal disorders) | 1 (1) — grade 3 mucositis
Nausea (Gastrointestinal disorders) | 1 (1) — grade 3 nausea
Pain - Abdomen NOS (General disorders) | 1 (1) — grade 3 pain
Pain - Head/headache (General disorders) | 1 (1) — grade 3 headache
weight loss (General disorders) | 2 (2) — grade 3 weight loss
anorexia (Gastrointestinal disorders) | 1 (1) — grade 3 anorexia
low CD4 count (Blood and lymphatic system disorders) | 1 (1) — grade 3 decrease in CD4 counts
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study (N=17)
Rhinitis (Immune system disorders) | 1 (1) — grade 1 rhinitis: 1 patient
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) — Lymphopenia in 5 patients (1 grade 1, 3 grade 2, 1 grade 3), not including the 2 patients with lymphopenia SAEs.
Hypertension (Cardiac disorders) | 1 (1) — Hypertension, 1 grade 2. This is in addition to the 1 grade 3 SAE.
Fatigue (General disorders) | 11 (11) — 6 grade 1, 5 grade 2.
Pruritis/itching (Skin and subcutaneous tissue disorders) | 8 (8) — 6 grade 1 , 2 grade 2
Mucositis - funct/sympt oral (Gastrointestinal disorders) | 7 (7) — 4 grade 1, 3 grade 2, in addition to 1 grade 3 SAE
Hemorrhage / Bleeding (Blood and lymphatic system disorders) | 8 (8) — 7 grade 1, 1 grade 2.
Infection, normal ANC, abdomen (Infections and infestations) | 1 (1) — 1 grade 2.
Edema - limb (Blood and lymphatic system disorders) | 4 (4) — Edema: 1 grade 1, 2 grade 2
Nausea (Gastrointestinal disorders) | 9 (9) — 7 grade 1, 2 grade 2, in addition to the one grade 3 SAE.
Urinary frequency (Renal and urinary disorders) | 1 (1) — one grade 1 urinary frequency
Hypotension (Cardiac disorders) | 4 (4) — hypotension: 3 grade 1, 1 grade 2
Fever (General disorders) | 6 (6) — Fever: 3 grade 1, 3 grade 2
Rigors/chills (General disorders) | 9 (9) — 8 grade 1, 1 grade 2
Sweating (General disorders) | 1 (1) — 1 grade 1.
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13 (13) — rash: 12 grade 1, 1 grade 2.
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2) — 1 grade 1, 1 grade 2
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12) — 12 grade 1 only.
Rash - acneiform (Skin and subcutaneous tissue disorders) | 6 (6) — 6 grade 1 only.
Wound complications, non-infectious (Skin and subcutaneous tissue disorders) | 4 (4) — 4 grade 1.
Hair loss / alopecia (Skin and subcutaneous tissue disorders) | 3 (3) — 3 grade 1.
Dermatology - other (Skin and subcutaneous tissue disorders) | 1 (1) — 1 grade 1.
Weight loss (General disorders) | 9 (9) — 4 grade 1, 5 grade 2, plus 2 wt loss SAEs.
Anorexia (Gastrointestinal disorders) | 12 (12) — 10 grade 1, 2 grade 2, in addition to 1 grade 3 SAE.
vomiting (Gastrointestinal disorders) | 5 (5) — 4 grade 1, 1 grade 1
mucositis - larynx (Gastrointestinal disorders) | 3 (3) — 3 grade 1
dry mouth (Gastrointestinal disorders) | 2 (2) — 2 grade 1
mucositis - esophagus (Gastrointestinal disorders) | 1 (1) — 1 grade 1.
colitis (Gastrointestinal disorders) | 1 (1) — 1 grade 1
dehydration (Gastrointestinal disorders) | 1 (1) — 1 grade 1
GI - other (Gastrointestinal disorders) | 1 (1) — 1 grade 1
Hemorrhage - lung (Blood and lymphatic system disorders) | 1 (1) — 1 grade 1
Hemorrhage - rectal (Blood and lymphatic system disorders) | 1 (1) — 1 grade 1
Infection, normal ANC, oral cavity (Infections and infestations) | 1 (1) — 1 grade 2
Infection (other) (Infections and infestations) | 1 (1) — 1 grade 1
Edema - head and neck (Blood and lymphatic system disorders) | 1 (1) — 1 grade 1
Hypophosphatemia (Investigations) | 3 (3) — 3 grade 2, in addition to 2 grade 3 (SAE)
Hypokalemia (Investigations) | 3 (3) — 3 grade 1, in addition to 2 grade 3 SAEs
Proteinuria (Investigations) | 7 (7) — 4 grade 1, 3 grade 2.
hypertriglyceridemia (Investigations) | 9 (9) — 8 grade 1, 1 grade 2
AST (Investigations) | 8 (8) — Elevated AST: 7 grade 1, 1 grade 2.
Alkaline phosphatase (Investigations) | 5 (5) — Elevated alkaline phosphatase: 4 grade 1, 1 grade 2.
Bilirubin (Investigations) | 4 (4) — 3 grade 1, 1 grade 2
Creatinine (Investigations) | 3 (3) — Elevated creatinine: 2 grade 1, 1 grade 2
Hypoalbuminemia (Investigations) | 2 (2) — 1 grade 1, 1 grade 2
Cholesterol (Investigations) | 10 (10) — Increased cholesterol: 10 grade 1
low serum bicarbonate (Investigations) | 7 (7) — grade 1: 7
ALT (Investigations) | 4 (4) — Elevated ALT: 4 grade 1
hyponatremia (Investigations) | 2 (2) — 2 grade 1.
acidosis (Investigations) | 1 (1) — 1 grade 1
hemoglobinuria (Investigations) | 1 (1) — 1 grade 1
hypercalcemia (Investigations) | 1 (1) — 1 grade 1
hypernatremia (Investigations) | 1 (1) — 1 grade 1
hypomagnesemia (Investigations) | 1 (1) — 1 grade 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) — 3 grade 1, 1 grade 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 2
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 1
Pain - extremity (Musculoskeletal and connective tissue disorders) | 2 (2) — 2 grade 1
Pain - joint (Musculoskeletal and connective tissue disorders) | 2 (2) — 2 grade 1
Pain - muscle (Musculoskeletal and connective tissue disorders) | 2 (2) — 2 grade 1
Pain - oral cavity (Respiratory, thoracic and mediastinal disorders) | 2 (2) — 2 grade 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — 2 grade 1
Pain - chest wall (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 1
Pain - oral - gums (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 1
Pain - other (General disorders) | 1 (1) — 1 grade 1
Pain - scalp (Skin and subcutaneous tissue disorders) | 1 (1) — 1 grade 1
Pain - skin (Skin and subcutaneous tissue disorders) | 1 (1) — 1 grade 1
pain - throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 1
Urinary frequency (Renal and urinary disorders) | 1 (1) — 1 grade 1
flu-like syndrome (General disorders) | 1 (1) — 1 grade 1
Pain - anus (Gastrointestinal disorders) | 1 (1) — 1 grade 2
Pain - stomach (Gastrointestinal disorders) | 1 (1) — 1 grade 2
Pain - tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — 1 grade 2
Pain - abdomen NOS (Gastrointestinal disorders) | 3 (3) — 2 grade 1, 1 grade 2, in addition to the one grade 3 SAE
Pain - headache (Nervous system disorders) | 7 (7) — seven grade 1, in addition to the one grade 3 SAE.
hemoglobin (Blood and lymphatic system disorders) | 13 (13) — low hemoglobin: 8 grade 1, 5 grade 2, in addition to the one grade 3 SAE
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 14 (14) — 11 grade 1, 3 grade 2
Hyperglycemia (Endocrine disorders) | 8 (8) — 3 grade 1, 5 grade 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — 1 grade 1, muscle weakness, lower extremity
Diarrhea (Gastrointestinal disorders) | 10 (10) — 6 grade 1, 4 grade 2
mucositis - clinical exam - oral (Gastrointestinal disorders) | 10 (10) — 7 grade 1, 3 grade 2
Leukocytes (Blood and lymphatic system disorders) | 6 (6) — 4 grade 1, 2 grade 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) — 5 grade 1, 1 grade 2
Neutrophils (Blood and lymphatic system disorders) | 4 (4) — 3 grade 1, 1 grade 2
Neuropathy - sensory (Nervous system disorders) | 3 (3) — 2 grade 1, 1 grade 2
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) — 1 grade 2
mucositis - vaginal (Reproductive system and breast disorders) | 1 (1) — 1 grade 2
taste alteration (Gastrointestinal disorders) | 10 (10) — 10 grade 1
constipation (Gastrointestinal disorders) | 6 (6) — 6 grade 1
voice changes (General disorders) | 6 (6) — 6 grade 1
Hypocalcemia (Investigations) | 4 (4) — 4 grade 1
nasal/paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 3 (3) — 3 grade 1
cognitive disturbance (Nervous system disorders) | 2 (2) — 2 grade 1
Dizziness (Ear and labyrinth disorders) | 2 (2) — 2 grade 1
Heartburn (Gastrointestinal disorders) | 2 (2) — 2 grade 1
hypopigmentation - skin (Skin and subcutaneous tissue disorders) | 1 (1) — 1 grade 1
urticaria (Skin and subcutaneous tissue disorders) | 1 (1) — 1 grade 1
Confusion (Nervous system disorders) | 1 (1) — 1 grade 1
Memory impairment (Nervous system disorders) | 1 (1) — 1 grade 1
Mood alteration - anxiety (Nervous system disorders) | 1 (1) — 1 grade 1
Tremor (Nervous system disorders) | 1 (1) — 1 grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less